CLINICAL TRIAL: NCT01392937
Title: The Clinical Performance of the All-in-One Light Multi-purpose Care Regimen for Silicone Hydrogel Contact Lenses
Brief Title: Clinical Performance of All-in-One Light Multi-purpose for Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sauflon Pharmaceuticals Ltd (Industry)
Responsible Party: Howard Griffiths, Sauflon Pharmaceuticals Limited
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: S09-469
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: AIOL; multipurpose solution; silicone hydrogel lenses; The safety and efficacy of the All-in-One Light multipurpose care regimen by comparison with the Aquify care regimen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- All-in-One Light multipurpose (Active Comparator): Used All in One light multipurpose with one of five different lens brands: Air Optix Aqua(Ciba Vision Inc.), PureVision (Bausch + Lomb Inc.), Biofinity (CooperVision Inc.), Acuvue Advance and Acuvue 2 (both Johnson & Johnson).
  Interventions: Device: All-in-One Light multipurpose
- Aquify care (Active Comparator): Use Aquify care with one of five different lens brands: Air Optix Aqua(Ciba Vision Inc.), PureVision (Bausch + Lomb Inc.), Biofinity (CooperVision Inc.), Acuvue Advance and Acuvue 2 (both Johnson & Johnson).
  Interventions: Device: Aquify care

INTERVENTIONS:
Device: All-in-One Light multipurpose — The study was conducted over two months of wear. Subjects were examined initially, and at three follow-up visits after two weeks, one month and two months.
  Arms: All-in-One Light multipurpose
Device: Aquify care — The study was conducted over two months of wear. Subjects were examined initially, and at three follow-up visits after two weeks, one month and two months.
  Arms: Aquify care

SUMMARY:
A clinical trial was conducted to assess the safety and acceptability of the Sauflon Multipurpose Solution when used with four different silicone hydrogel contact lens brands and one conventional hydrogel control lens was conducted over a period of two months, with a control group using Ciba Vision Aquify Multi- Purpose Solution. The study was conducted at six investigator sites and a total of 257 subjects were enrolled. The results of this study showed the safety, acceptability and substantial equivalence of the Sauflon Multipurpose Solution to the predicate device for its intended use.

DETAILED DESCRIPTION:
1.1 Study characteristics This study evaluated the safety and efficacy of the All-in-One Light multipurpose care regimen (Sauflon Pharmaceuticals Limited) by comparison with the Aquify care regimen(Ciba Vision Inc.). Each subject used one of five different lens brands: Air Optix Aqua(Ciba Vision Inc.), PureVision (Bausch + Lomb Inc.), Biofinity (CooperVision Inc.), Acuvue Advance and Acuvue 2 (both Johnson & Johnson).

The key study features were as follows:

1. Two months duration.
2. Six investigator sites.
3. Daily wear soft (hydrophilic) contact lenses, replaced on a two-weekly basis: Air Optix Aqua, PureVision, Biofinity, Acuvue Advance and Acuvue 2; with one of two care regimens: All-in-One Light and Aquify.
4. A total of 257 subjects were enrolled, and 256 subjects accounting for 512 eyes were dispensed lenses. This group was randomized into 173 test subjects (346 eyes) and 83 control subjects (166 eyes).
5. Of the 173 test subjects, 163 (94.2%) completed two months of use. Of the 83 control subjects, 73 (88.0%) completed two months of use.
6. No eyes remained active at the end of the study.
7. There were no adverse reactions. 1.2 Study period The study was conducted over two months of wear. Subjects were examined initially, and at three follow-up visits after two weeks, one month and two months. Study visits commenced on March 29, 2010 and were completed on March 11, 2011.

1.3 Demographics Six investigator sites dispensed 173 test subjects (346 eyes) who used All-in-One Light as their care regimen during the work. Also dispensed were 83 control subjects (166 eyes)who used Aquify as their care regimen during the work. All recruited subjects were existing contact lenses wearers.

Of the 173 test subjects, 163 (94.2%) completed two months of use and ten (5.8%) were discontinued. Of the 83 control subjects, 73 (88.0%) completed two months of use and ten (12.2%) were discontinued.

The enrolled control group was made up of 51 females (61%) and 32 males (39%) with an age range from 18 to 67 years (mean 36.7 years). The enrolled test group was composed of 117 females (67%) and 57 males (33%) with an age range from 18 to 65 years (mean 34.1 years). One subject (female, age 45 years) was enrolled and assigned to the test group but was not dispensed lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They are 18 years of age and above.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research for the duration of this study.
  5. They can attain at least 6/12 in each eye with the study contact lenses.
  6. They have successfully worn contact lenses within six months of starting the study.
  7. They can be fitted with spherical soft contact lenses within the power ranges of the study lenses.

Exclusion Criteria:

* Subjects will not be eligible if:

  1. They have an ocular disorder which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They are aphakic.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
  7. They are pregnant or lactating.
  8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
  9. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall subjective acceptance. | 2 months
  The safety and efficacy of the All-in-One Light multipurpose care regimen (Sauflon Pharmaceuticals Limited) by comparison with the Aquify care regimen(Ciba Vision Inc.). Each subject used one of five different lens brands: Air Optix Aqua(Ciba Vision Inc.), PureVision (Bausch + Lomb Inc.), Biofinity (CooperVision Inc.), Acuvue Advance and Acuvue 2 (both Johnson & Johnson).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, Principal Investigator — MCOptom FAAO FBCLA
Locations (1):
- Eurolens Research Faculty of Life Sciences The University of Manchester, Manchester, Manchester, United Kingdom